CLINICAL TRIAL: NCT04205344
Title: Effectiveness of Subarachnoid Hyperbaric Bupivacaine on Mean Arterial Blood Pressure in Pregnant Patients With Obesity Operated by Cesarean Section
Brief Title: Subarachnoid Bupivacaine in Obese Patients Undergoing Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, MARIA DE LOS ANGELES CAMPECHANO ASCENCIO, Anesthesiologist, Hospital Civil de Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 005/16
Record Dates: First submitted 2019-12-07; First posted 2019-12-19 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Anesthesia, Obstetrical
Keywords: Bupivacaine; Obesity; Pregnant; Subarachnoid; Cesarean; Subdural
MeSH Terms: conditions — Obesity | interventions — Bupivacaine; Glucose

STUDY DESIGN:
Intervention Model Description: Clinical trial open controlled parallel randomized simple
Who Masked: Participant, Investigator
Masking Description: You do not know the dose of bupivacaine you receive
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupivacaine 5 mg (Experimental): Receive subarachnoid hyperbaric bupivacaine at a dose of 5 mg
  Interventions: Drug: Bupivacaine 5 mg
- Bupivacaine 10 mg (Experimental): Receive subarachnoid hyperbaric bupivacaine at a dose of 10 mg
  Interventions: Drug: Bupivacaine 10 mg

INTERVENTIONS:
Drug: Bupivacaine 5 mg — Receive subarachnoid hyperbaric bupivacaine at a dose of 5 mg
  Other Names: hyperbaric bupivacaine 1ml; bupivacaine/Dextrose 1ml
  Arms: Bupivacaine 5 mg
Drug: Bupivacaine 10 mg — Receive subarachnoid hyperbaric bupivacaine at a dose of 10 mg
  Other Names: hyperbaric bupivacaine 2 ml; bupivacaine/Dextrose 1 ml
  Arms: Bupivacaine 10 mg

SUMMARY:
This study evaluates the effect of subarachnoid hyperbaric bupivacaine on mean arterial blood pressure (MAP) of pregnant patients with obesity undergoing cesarean section half of the patients will receive subarachnoid hyperbaric bupivacaine at a dose of 5 mg while the other half will receive a dose of 10 mg

DETAILED DESCRIPTION:
Once the patients were admitted to the toco-surgery work area, patients over 18 years of age were captured, with pregnancy ≥37 weeks of gestation, which, based on weight and height prior to pregnancy, obesity is diagnosed with a BMI ≥30 kg / m2 and that had an indication of termination of pregnancy via abdominal caesarean section without compromising fetal well-being. Specifically, the objectives of the study protocol, benefits and risks were given and it was given to choose an envelope containing the consent letter under information, the data collection sheet and the group to which it was assigned. He was granted the consent letter under information to sign; the same procedure was performed with the husband or relative responsible for the patient They underwent pre-anesthetic evaluation, background check and review of laboratory tests, as well as taking vital signs such as non-invasive blood pressure, mean blood pressure (PAM), O2 saturation and heart rate, Fetal heart rate was taken with adult stethoscope. The administration of Hartmann solution at 10ml /kg pregestational weight and premedication with ranitidine 50 mg and metoclopramide 10 mg was informed prior to admission to the operating room In the operating room, room preparation was carried out with material for anesthesiology corresponding laryngoscope, intubation cannulas, oropharyngeal cannulas, verification of operation of anesthesia machine, verification of material of blocking equipment, needles, syringes, alcohol and iodo povidone; Verify hyperbaric bupivacaine drugs, ephedrine and atropine. In case of requiring a change in anesthetic technique, general anesthesia have necessary fentanyl opioid drugs, propofol inducer and rocuronium muscle relaxant. Preparation of emergency drugs atropine and ephedrine dilution of 1 ampoule in 10 ml of diluent solution. The patient was transferred to the operating room, baseline vital signs were taken, non-invasive blood pressure, MAP, O2 saturation and heart rate with the monitor team Simultaneously fetal heart rate was taken Permeability of peripheral pathways was verified The patient was placed in a sitting position and started with mixed technique neuraxial anesthetic anesthetic technique (placement of peridural catheter + subarachnoid block with brand blocking equipment) The anatomical reference of the intervertebral space L2-L3, L3-L4 was located in a seated position. Aseptic and antiseptic technique was performed with iodo povidone, and subsequently removed with alcohol Sterile fields were placed Skin and subcutaneous tissue were infiltrated with 2% lidocaine 5 ml of the selected intervertebral space Tuohy needle No. 17 was introduced with the "Gout of Gutierrez" technique, until the location was found, it was corroborated with the "resistance loss" technique. Through the Tuohy needle, the spinal needle "whitacre" pencil No. 27 was introduced until cerebrospinal fluid (CSF) was obtained. The dose of hyperbaric bupivacaine blockade of 10 mg (2 ml) or mg (1 ml) was administered agreement with the assigned group, in approximately 20 seconds; the spinal needle pencil tip "whitacre" and an epidural catheter was introduced with cephalic direction and left 5 cm inside the epidural space, left inert. Catheter was attached to the back with adhesive tape The patient was placed in a dorsal recumbent position with a shifting wedge placement on the right hip approximately 15 degrees to the left. Vital signs monitoring was started every 3 minutes for the first 15 minutes and then every 5 minutes until the end of the anesthetic procedure When obtaining PAM record of less than 20% at baseline, ephedrine 10 mg is administered and total doses required were recorded until PAM records were recovered above 20% of baseline. Together with the record of the first taking of vital signs, the fetal heart rate was taken again After the second vital signs were taken, (3 minutes), a sensory block evaluation was started with a puncture technique from the dermatome where the block was placed and the ascending dermatome was registered where the patient reported pain. This assessment was performed every 3 minutes for the first 15 minutes, and then every 15 minutes until the end of the surgery. The blocking level was considered adequate to initiate the surgical procedure when the loss of sensitivity in the T4 dermatome was reached. After the second vital signs were taken (3 minutes), a motor block assessment with a Bromage scale was initiated, in which the patient was instructed to make movements with her legs to assess the capacity of movement that still remains. This assessment was performed every 3 minutes for the first 15 minutes, and then every 15 minutes until the end of the surgery After the second vital signs were taken (3 minutes), the patient was asked if she had a feeling of nausea or the presence of vomiting and was registered. At the extraction of the fetus, the Apgar assessment granted by the attached neonatology doctor at one minute and at 5 minutes of extrauterine life was recorded. Once the placenta was illuminated, a sample was taken for gasometry with a heparinized syringe of the umbilical artery and sent to the laboratory for processing. A dose of local anesthetic was administered via a 5% lidocaine 2% peridural catheter if necessary, when the patient reported discomfort or pain (referred to the decrease in sensory block) and the surgical procedure has not been completed. The time at which subsequent doses are administered is recorded The information collected was recorded on the data collection sheet. The presence of adverse reactions to drugs or the anesthetic technique were recorded in the adverse event sheets. The sample size was calculated with a formula for comparison of two means with finite population.

No results are found in previous publications with a statistically significant P, so a pilot test is carried out based on the specified criteria, which includes 30 patients, 15 patients in the group administered 5 mg of Subarachnoid hyperbaric bupivacaine and 15 patients in the group who were administered 10 mg of the same drug, and a standard deviation of 14.46 was obtained for the maximum blood hypotension variable recorded. For the development of the finite population formula, the total of anesthesiology procedures is quantified, the total of cesarean surgeries performed in the operating rooms of the toco-surgery of the Civil Hospital of Guadalajara Fray Antonio Alcalde in 2015; where a total of 1,218 caesarean sections are obtained y Calculated losses 25% pregnant women with obesity per group N = 40 patients. The statistical analysis was carried out once both study groups were completed. The groups were divided with the assignment codes to group 5 or 10. The database was formed in the Microsoft Office Excel 2013 program, which was exported to the statistical program Statistics Product and Service Solution (SPSS) version 22 in order to carry out the data analysis. All patients were included in the statistical analysis. The data obtained are expressed through measures of central tendency and dispersion, mean and standard deviation for quantitative variables, and frequencies and percentages in the case of qualitative variables. Due to the sample size, it is decided to use non-parametric tests for data analysis. The intra-group differences for the quantitative variables were determined by the Wilcoxon rank test, while the differences between the groups were determined with the Mann Whitney U test. Qualitative variables were analyzed through the Chi Square test. A value of p≤0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with single fetus pregnancy ≥37 weeks gestation
* Body mass index (BMI) ≥ 30 kg / m2
* Indication of termination of pregnancy via abdominal caesarean section
* Indication of subarachnoid neuraxial block under mixed technique
* Signing of consent under information

Exclusion Criteria:

* Patients with a known allergy to local anesthetics
* Patients with psychiatric treatment (antidepressants, anxiolytics, antipsychotics)
* Patients with addiction to any type of drug
* Patients with a history of liver disease
* Patients with a history of renal pathology
* Patients with a history of pulmonary pathology
* Patients with a history of cardiac pathology
* Patients with a history of high blood pressure
* Patient with a history of type I, II and gestational diabetes
* Non-calming fetal state
* Patients who refuse the anesthetic technique of neuraxial block

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — single fetus pregnancy whit BMI≥ 30 kg/m2
Enrollment: 40 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Assess the mean blood pressure | 2 hours
  Number of participants with a decrease in mean arterial blood pressure after administration of subarachnoid hyperbaric bupivacaine at a dose of 5 mg and 10 mg to preserve the mean blood pressure in pregnant patients with obesity undergoing caesarean section
Determine the effects on the heart rate | 2 hour
  Number of participants presenting changes in heart rate such as bradycardia (heart rate less than 60 beats minute) or tachycardia (heart rate greater than 120 beats minute) after administration of subarachnoid hyperbaric bupivacaine in the pregnant patients with obesity, after subarachnoid block
Determine the effects on the respiratory rate | 2 hour
  Number of participants presenting changes in respiratory rate such as bradypnea (respiratory rate less than 12 minute breaths) after administration of subarachnoid hyperbaric bupivacaine in the pregnant patient with obesity, after subarachnoid block

SECONDARY OUTCOMES:
Describe the adverse effects | 2 hours
  Number of participants with side effects such as nausea or vomiting after administration of subarachnoid hyperbaric bupivacaine in the pregnant patient with obesity, after subarachnoid block.
Identify the level of sensory blockade | 15 minutes
  The number of participants with adequate sensory block (thoracic dermatome 4 is defined as adequate to begin the surgical technique), the level of sensory block reached after the subarachnoid block; The sensory block was evaluated using pinprick. Every 3 minutes the first 15 minutes after the subarcnoid block.
Identify the intensity of motor blockade | 15 minutes
  The number of participants with adequate intensity of motor blockade achieved after subarachnoid block, the intensity of the motor block was evaluated with the bromage scale (I Free movement of legs and feet. II Just able to flex Knees with free movement of feet, III Unable to flex knees, but with free movement of feet. IV Unable to move legs or feet) Level IV was considered adequate motor block. Every 3 minutes the first 15 minutes after the subarachnoid block.
Measure the duration of the block | 2 hour
  Measure the duration of the block with a dose of 5 mg and 10 mg of hyperbaric bupivacaine via subarachnoid route in pregnant patients with obesity
Describe the adverse effects on the fetus | 1 hour
  The number of patients with any side effect associated with the fetal bradycardia anesthetic technique (Fetal heart rate less than 120 beats minute) cardiac arrest (Fetal heart rate less than 100 beats minute) And in the newborn fetal acidosis (umbilical vein gasometry with Hydrogen Potential (pH) <7.0 or excess bases >-12 mmol/L)
Document the Apgar score | 5 minutes
  Document the Apgar score in the newborn. (Apgar Score evaluate five sign: color, heart rate, reflex irritability, muscle tone and respiration) The score ranges from 0 to 2 per sign according to the criteria of the neonatologist, to grant a maximum score of 10 points. A grade of less than 7 points is considered low Apgar scores. This scores is registered t minute and five minutes of life.

CONTACTS AND LOCATIONS:
Overall Officials: MARIA DE LOS ANGELES CAMPECHANO ASCENCIO, MSc, Principal Investigator — Hospital Civil de Guadalajara; MIRIAM MENDEZ DEL VILLAR, MSc PhD, Study Director — CENTRO UNIVERSITARIO DE TONALA; LEONEL GARCIA BENAVIDES, Study Chair — Hospital Civil de Guadalajara; JORGE BRAVO RUBIO, Study Chair — Hospital Civil de Guadalajara
Locations (1):
- Hospital Civil de Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teoh WH, Thomas E, Tan HM. Ultra-low dose combined spinal-epidural anesthesia with intrathecal bupivacaine 3.75 mg for cesarean delivery: a randomized controlled trial. Int J Obstet Anesth. 2006 Oct;15(4):273-8. doi: 10.1016/j.ijoa.2006.03.004. Epub 2006 Jun 13. PMID 16774830
- [Result] Tonidandel A, Booth J, D'Angelo R, Harris L, Tonidandel S. Anesthetic and obstetric outcomes in morbidly obese parturients: a 20-year follow-up retrospective cohort study. Int J Obstet Anesth. 2014 Nov;23(4):357-64. doi: 10.1016/j.ijoa.2014.05.004. Epub 2014 Jun 4. PMID 25201313
- [Result] Ouzounian JG, Elkayam U. Physiologic changes during normal pregnancy and delivery. Cardiol Clin. 2012 Aug;30(3):317-29. doi: 10.1016/j.ccl.2012.05.004. Epub 2012 Jun 20. PMID 22813360
- [Result] Hood DD, Dewan DM. Anesthetic and obstetric outcome in morbidly obese parturients. Anesthesiology. 1993 Dec;79(6):1210-8. doi: 10.1097/00000542-199312000-00011. PMID 8267196
- [Result] Tan T, Sia AT. Anesthesia considerations in the obese gravida. Semin Perinatol. 2011 Dec;35(6):350-5. doi: 10.1053/j.semperi.2011.05.021. PMID 22108086
- [Result] Ngan Kee WD, Khaw KS, Tan PE, Ng FF, Karmakar MK. Placental transfer and fetal metabolic effects of phenylephrine and ephedrine during spinal anesthesia for cesarean delivery. Anesthesiology. 2009 Sep;111(3):506-12. doi: 10.1097/ALN.0b013e3181b160a3. PMID 19672175
- [Result] Lee Y, Balki M, Parkes R, Carvalho JC. Dose requirement of intrathecal bupivacaine for cesarean delivery is similar in obese and normal weight women. Rev Bras Anestesiol. 2009 Nov-Dec;59(6):674-83. doi: 10.1016/s0034-7094(09)70092-3. English, Portuguese. PMID 20011857
- [Result] Carvalho B, Collins J, Drover DR, Atkinson Ralls L, Riley ET. ED(50) and ED(95) of intrathecal bupivacaine in morbidly obese patients undergoing cesarean delivery. Anesthesiology. 2011 Mar;114(3):529-35. doi: 10.1097/ALN.0b013e318209a92d. PMID 21307769
- [Result] Ring LE. The anesthetic approach to operative delivery of the extremely obese parturient. Semin Perinatol. 2014 Oct;38(6):341-8. doi: 10.1053/j.semperi.2014.07.008. Epub 2014 Aug 19. PMID 25146109
- [Result] Badve MH, Golfeiz C, Vallejo MC. Anesthetic considerations for the morbid obese parturient. Int Anesthesiol Clin. 2014 Summer;52(3):132-47. doi: 10.1097/AIA.0000000000000024. No abstract available. PMID 24946047
- [Result] Lamon AM, Habib AS. Managing anesthesia for cesarean section in obese patients: current perspectives. Local Reg Anesth. 2016 Aug 16;9:45-57. doi: 10.2147/LRA.S64279. eCollection 2016. PMID 27574464
- [Result] Dennis AT, Castro JM, Ong M, Carr C. Haemodynamics in obese pregnant women. Int J Obstet Anesth. 2012 Apr;21(2):129-34. doi: 10.1016/j.ijoa.2011.11.007. Epub 2012 Feb 11. PMID 22326199
- [Result] Rodrigues FR, Brandao MJ. Regional anesthesia for cesarean section in obese pregnant women: a retrospective study. Rev Bras Anestesiol. 2011 Jan-Feb;61(1):13-20. doi: 10.1016/S0034-7094(11)70002-2. PMID 21334503
- [Result] Wise RA, Polito AJ, Krishnan V. Respiratory physiologic changes in pregnancy. Immunol Allergy Clin North Am. 2006 Feb;26(1):1-12. doi: 10.1016/j.iac.2005.10.004. PMID 16443140
- [Result] Chandra S, Tripathi AK, Mishra S, Amzarul M, Vaish AK. Physiological changes in hematological parameters during pregnancy. Indian J Hematol Blood Transfus. 2012 Sep;28(3):144-6. doi: 10.1007/s12288-012-0175-6. Epub 2012 Jul 15. PMID 23997449
- [Result] American College of Obstetricians and Gynecologists. ACOG Committee opinion no. 549: obesity in pregnancy. Obstet Gynecol. 2013 Jan;121(1):213-7. doi: 10.1097/01.aog.0000425667.10377.60. PMID 23262963
- [Result] Soens MA, Birnbach DJ, Ranasinghe JS, van Zundert A. Obstetric anesthesia for the obese and morbidly obese patient: an ounce of prevention is worth more than a pound of treatment. Acta Anaesthesiol Scand. 2008 Jan;52(1):6-19. doi: 10.1111/j.1399-6576.2007.01483.x. PMID 18173431
- [Result] Gaiser R. Anesthetic Considerations in the Obese Parturient. Clin Obstet Gynecol. 2016 Mar;59(1):193-203. doi: 10.1097/GRF.0000000000000180. PMID 26694495
- [Result] Nani FS, Torres ML. Correlation between the body mass index (BMI) of pregnant women and the development of hypotension after spinal anesthesia for cesarean section. Rev Bras Anestesiol. 2011 Jan-Feb;61(1):21-30. doi: 10.1016/S0034-7094(11)70003-4. PMID 21334504
- [Result] Klohr S, Roth R, Hofmann T, Rossaint R, Heesen M. Definitions of hypotension after spinal anaesthesia for caesarean section: literature search and application to parturients. Acta Anaesthesiol Scand. 2010 Sep;54(8):909-21. doi: 10.1111/j.1399-6576.2010.02239.x. Epub 2010 Apr 23. PMID 20455872
- [Result] Rasolonjatovo TY, Ravololonirina BM, Randriamanantany ZA, Raveloson NE. [Spinal anesthesia for cesarean section: risk factors for emergence of Apgar scores below 7 in Malagasy newborns]. Pan Afr Med J. 2014 Oct 23;19:193. doi: 10.11604/pamj.2014.19.193.3392. eCollection 2014. French. PMID 25821536
- [Result] Mercier FJ, Auge M, Hoffmann C, Fischer C, Le Gouez A. Maternal hypotension during spinal anesthesia for caesarean delivery. Minerva Anestesiol. 2013 Jan;79(1):62-73. Epub 2012 Nov 18. PMID 23135692
- [Result] Polin CM, Hale B, Mauritz AA, Habib AS, Jones CA, Strouch ZY, Dominguez JE. Anesthetic management of super-morbidly obese parturients for cesarean delivery with a double neuraxial catheter technique: a case series. Int J Obstet Anesth. 2015 Aug;24(3):276-80. doi: 10.1016/j.ijoa.2015.04.001. Epub 2015 Apr 8. PMID 25936783
- [Result] Sng BL, Siddiqui FJ, Leong WL, Assam PN, Chan ES, Tan KH, Sia AT. Hyperbaric versus isobaric bupivacaine for spinal anaesthesia for caesarean section. Cochrane Database Syst Rev. 2016 Sep 15;9(9):CD005143. doi: 10.1002/14651858.CD005143.pub3. PMID 27629425
- [Result] Eltzschig HK, Lieberman ES, Camann WR. Regional anesthesia and analgesia for labor and delivery. N Engl J Med. 2003 Jan 23;348(4):319-32. doi: 10.1056/NEJMra021276. No abstract available. PMID 12540646
- [Result] Hollowell J, Pillas D, Rowe R, Linsell L, Knight M, Brocklehurst P. The impact of maternal obesity on intrapartum outcomes in otherwise low risk women: secondary analysis of the Birthplace national prospective cohort study. BJOG. 2014 Feb;121(3):343-55. doi: 10.1111/1471-0528.12437. Epub 2013 Sep 11. PMID 24034832
- [Result] Zhu T, Tang J, Zhao F, Qu Y, Mu D. Association between maternal obesity and offspring Apgar score or cord pH: a systematic review and meta-analysis. Sci Rep. 2015 Dec 22;5:18386. doi: 10.1038/srep18386. PMID 26692415
- [Result] Edwards RK, Cantu J, Cliver S, Biggio JR Jr, Owen J, Tita ATN. The association of maternal obesity with fetal pH and base deficit at cesarean delivery. Obstet Gynecol. 2013 Aug;122(2 Pt 1):262-267. doi: 10.1097/AOG.0b013e31829b1e62. PMID 23969793
- [Result] Reyes M, Pan PH. Very low-dose spinal anesthesia for cesarean section in a morbidly obese preeclamptic patient and its potential implications. Int J Obstet Anesth. 2004 Apr;13(2):99-102. doi: 10.1016/j.ijoa.2003.09.004. PMID 15321413
- [Result] Bamgbade OA, Khalaf WM, Ajai O, Sharma R, Chidambaram V, Madhavan G. Obstetric anaesthesia outcome in obese and non-obese parturients undergoing caesarean delivery: an observational study. Int J Obstet Anesth. 2009 Jul;18(3):221-5. doi: 10.1016/j.ijoa.2008.07.013. Epub 2009 May 17. PMID 19447599
- [Result] Ngaka TC, Coetzee JF, Dyer RA. The Influence of Body Mass Index on Sensorimotor Block and Vasopressor Requirement During Spinal Anesthesia for Elective Cesarean Delivery. Anesth Analg. 2016 Dec;123(6):1527-1534. doi: 10.1213/ANE.0000000000001568. PMID 27870737
- See also: Legislative power — http://www.diputados.gob.mx/LeyesBiblio/regley/Reg_LGS_MIS.pdf
- See also: World Health Organization. Obesity and Overweight Descriptive Note No. 311 — http://www.who.int/mediacentre/factsheets/fs311/es/